CLINICAL TRIAL: NCT01651247
Title: Blinded Retrospective Laboratory Evaluations to Assess the Serologic Response to Porcine Circovirus Type 1 (PCV-1) in the Serum of Infants Aged 2 and 6 Months and Toddlers Aged 4-6 Years Following Administration of GlaxoSmithKline (GSK) Biologicals' IPV-containing Vaccines
Brief Title: Assessment of the Serologic Response to Porcine Circovirus Type 1 (PCV-1) in the Serum of Infants and Toddlers, Following Administration of IPV (Inactivated Poliovirus Vaccine)-Containing Vaccines
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114535; 213503/048; 217744/085
Record Dates: First submitted 2012-07-12; First posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Presence of Materials From PCV-1
Keywords: Toddlers; Retrospective; Porcine circovirus type 1 (PCV-1); Infants; Laboratory evaluations; IPV

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum

GROUPS / COHORTS (2):
- Group A: Subjects received 3 doses of the combination DTaP-HepB-IPV vaccine or separately administered DTaP, HepB, and IPV vaccines at 2, 4, and 6 months of age, in a previous study (217744/085).
  Interventions: Procedure: Serum sample
- Group B: Subjects received a single dose of the combination DTaP-IPV vaccine or separately administered DTaP and IPV vaccines at 4-6 years of age, in a previous study (213503/048).
  Interventions: Procedure: Serum sample

INTERVENTIONS:
Procedure: Serum sample — Serum samples collected at pre-determined time points in previously completed studies (217744/085 and 213503/048) will be analysed to detect the presence of anti PCV-1 antibodies.

SUMMARY:
This study aims to analyse the serologic response to PCV-1 in the PEDIARIX® [GSK Biologicals' Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine] and KINRIX® (GSK Biologicals' Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed and Inactivated Poliovirus Vaccine) vaccine products. The samples have been collected at pre-determined time points from a subset of subjects who participated in selected studies [217744/085 and 213503/048] conducted in the United States.

DETAILED DESCRIPTION:
Serum samples from the previously conducted clinical trials (217744/085 and 213503/048) are used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled previously in randomized, open and multicentre studies [217744/085; 213503/048].
* Subjects aged 6 months to 6 years at last dose vaccinated with either DTaP-HepB-IPV vaccine or separately administered DTaP, HepB, and IPV vaccines or DTaP-IPV vaccine or separately administered DTaP and IPV vaccines.
* Subjects for whom sufficient residual volume of the pre and post vaccination blood samples is available.

Exclusion Criteria:

* Not Applicable

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants aged 2 and 6 months who were previously given a primary vaccination series consisting of a single dose of combination DTaP-HepB-IPV (PEDIARIX®) vaccine at 2, 4, and 6 months of age or separately administered DTaP (INFANRIX®), HepB (ENGERIX-B®), and IPV (Sanofi-Pasteur's IPOL) vaccines in the study 217744/085 and toddlers aged 4-6 years who were previously vaccinated with a single dose of either the combination DTaP-IPV (KINRIX®) vaccine or separately administered DTaP and IPV vaccines in the study 213503/048.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Presence of serum anti-PCV-1 antibody. | At Day 0 and post vaccination time points (up to 1 month after vaccination).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline